CLINICAL TRIAL: NCT01117688
Title: Ureteroscopy With and Without Safety Guidewire:. A Prospective, Randomized Study of the Results of Endoscopic Treatment of Urolithiasis.
Brief Title: Ureteroscopy With and Without Safety Guidewire
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn. Not enough time to go through with the study.
Sponsor: Helse-Bergen HF (Other)
Responsible Party: Øyvind Ulvik, Helse-Bergen HF, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102.09 (REK) - 3; 21835 (NSD) - 3 (Other: Norway: Norwegian Social Science Data Services); 102.09 (REK) - 3 (Other: The National Committees for Research Ethics in Norway)
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2011-06

CONDITIONS: Urolithiasis
Keywords: Ureteroscopy
MeSH Terms: conditions — Urolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B - without SGW (Active Comparator): Ureteroscopy without SGW in place.
  Interventions: Procedure: Ureteroscopy with and without safety guidewire
- A - with SGW (Active Comparator): Ureteroscopy with SGW in place.
  Interventions: Procedure: Ureteroscopy with and without safety guidewire

INTERVENTIONS:
Procedure: Ureteroscopy with and without safety guidewire — In study arm A - with SGW, endoscopic treatment is performed with a safety guidewire in place. In study arm B - without SGW, the ureteroscopy is performed without SGW.

SUMMARY:
The purpose of this study is to investigate the impact of a safety guidewire (SGW) on the results of ureteroscopy for urolithiasis.

Study hypothesis: Routine use of SGW has no impact on the results of ureteroscopic treatment of urolithiasis.

DETAILED DESCRIPTION:
The use of SGW is generally recommended at any ureteroscopic procedure in order to facilitate the introduction of the endoscope and to secure placement of internal tubes for drainage of urine after the procedure.

However, SGW may be an obstacle to efficient disintegration and retraction of calculi in the narrow ureter.

The intention of this study is to compare the results of endoscopic stone treatment with and without the use of SGW.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urolithiasis planned for ureterorenoscopic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Stone free-rate | 3 months after treatment

SECONDARY OUTCOMES:
Hospital stay | Up to 1 week after the operation
Complication rate | Until 3 months after the procedure
Operating time | Up to 1 day after the surgery

CONTACTS AND LOCATIONS:
Overall Officials: Øyvind Ulvik, MD, Principal Investigator — Helse Bergen HF, Haukeland University Hospital
Locations (1):
- Helse Bergen HF, Haukeland University Hospital, Bergen, Bergen, Norway